CLINICAL TRIAL: NCT01599208
Title: Facilitating Associative Memory Via Deep Transcranial Magnetic Stimulation to the Medial Temporal Lobe
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: no IRB
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TMS-MEMORY-1
Record Dates: First submitted 2012-05-07; First posted 2012-05-15 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Effect of Deep Transcranial Magnetic Stimulation on Memory

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Single-pulse online stimulation (Experimental): Online single-pulse online stimulation at 120% of motor threshold to either the right or left MTL, in comparison to sham condition, in either -400/0/400/800 ms relatively to stimulus in either the study or test phases of a recognition test.
  Interventions: Device: TMS
- Repetitive online stim., 400ms, 10Hz (Experimental): Repetitive online stimulation for 400ms at 10Hz at 120% of motor threshold to either the right or left MTL, in comparison to sham condition, in either -400/0/400/800 ms relatively to stimulus in either the study or test phases of a recognition test.
  Interventions: Device: TMS
- Repetitive online stim., 400ms, 20Hz (Experimental): Repetitive online stimulation for 400ms at 20Hz at 120% of motor threshold to either the right or left MTL, in comparison to sham condition, in either -400/0/400/800 ms relatively to stimulus in either the study or test phases of a recognition test.
  Interventions: Device: TMS
- Repetitive offline stimulation at 10Hz (Experimental): Repetitive offline stimulation at 10Hz for 4 min before study or for 8 min before test (in accordance with the phase length), comprising 2-second stimulation trains and 20-second breaks. Stimulation will be given at 120% of motor threshold to either the right or the left MTL in comparison to sham condition.
  Interventions: Device: TMS
- Repetitive offline stimulation at 20Hz (Experimental): Repetitive offline stimulation at 20Hz for 4 min before study or for 8 min before test (in accordance with the phase length), comprising 2-second stimulation trains and 20-second breaks. Stimulation will be given at 120% of motor threshold to either the right or the left MTL in comparison to sham condition.
  Interventions: Device: TMS
- Repetitive offline stimulation with iTBS (Experimental): Repetitive offline stimulation with Intermittent Theta Burst Stimulation (iTBS) comprising 3 pulses at 50Hz, repeated at 5Hz for 2-second stimulation trains with 8-second breaks for 192 seconds. Stimulation will be given at 90% of motor threshold to either the right or the left MTL in comparison to sham condition.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — TRANSCRANIAL MAGNETIC STIMULATION

SUMMARY:
The goal of the proposed research is to map the effects-in particular facilitation-of Transcranial Magnetic Stimulation (TMS) of the Medial Temporal Lobes (MTL) onto the processing of associative memory. TMS technology has the potential to selectively enhance functions mediated by areas in the temporal cortex, including the MTL, known to be the primary neuronal seat of episodic memory. By using this technology the investigators can further our understanding of theoretical models of human memory (specifically regarding the role of Recollection and Familiarity processes), and additionally, provide a possible route to the recovery of some of memory loss typically observed in the elderly-namely, memory for associations. Given the MTL's critical role in human memory and facilitation-inducing qualities of TMS, this research goal is to provide a nonintrusive tool to facilitate memory performance in young and elderly healthy participants.

DETAILED DESCRIPTION:
Our theoretical motivation is to explore the mechanisms underlying recognition memory. Evidence from a variety of paradigms has converged on the notion that recognition memory comprises two processes:

1. Familiarity, entails item-specific information.
2. Recollection, entails association-specific information. Evidence suggests that recollection is associated with a network of neuronal regions, including the anterior medial prefrontal cortex, lateral parietal cortex, and the hippocampus. Familiarity, in contrast, is associated with the lateral prefrontal cortex and the peripheral cortex. Critically, for both familiarity and recollection, the vital role of the MTL is strongly implicated. To dissociate between recollection and familiarity, despite stimulating the same location in the brain, the investigators take into account the difference in processing time in which these two processes are known to operate, and use both objective and subjective cognitive tasks to accurately measure effects.

In addition, this research has clinical motivation, which relates to the nature of memory decline in the elderly. If successful, the investigators will be able to set an effective TMS protocol that could be used as a tool to enhance the very types of memories-association-specific memories-that are thought to mediate poor memory performance in the elderly.

To achieve both goals, the proposed experiments will target the MTL using both online stimulation (short-duration stimulation during the presentation of stimuli in recognition memory test) that will enable us to differentiate between effects of familiarity and recollection and offline stimulation mode (repetitive stimulation of several minutes separately from the recognition memory test), with the goal of achieving facilitation effects on memory performance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-85
* Answered negatively on safety screening questionnaire for TMS
* Capable and willing to provide informed consent.
* For participants aged more than 65, normal memory scoring should be obtained in a Nexig test.

Exclusion Criteria:

* History of epilepsy or seizure or history of such in first degree relatives.
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure, or history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes.
* History of head injury necessitating cranial surgery or prolonged coma.
* History of any metal in the head including the eyes and ears (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* History of severe migraine.
* History of significant hearing loss.
* Individuals with a significant neurological disorder.
* History of substance abuse including alcoholism within the past 6 months (except nicotine and caffeine)
* Inadequate communication with the participant.
* Participation currently in another clinical study or enrolled in another clinical study within 30 days prior to this study.
* Participants who suffer from an unstable physical, systemic and metabolic disorders
* Women who are breast-feeding
* Known or suspected pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change in memory based on the timeframe of the online stimulation | One year
  For the online stimulation arms, we expect to find a change in memory based on the timeframe of the online stimulation and the cognitive task, namely, we expect to find change in memory for associations when stimulation is at around 800ms, and expect a change in memory for items when stimulation is at around 400ms.

CONTACTS AND LOCATIONS:
Overall Officials: Yonatan Goshen, Prof., Principal Investigator — Tel Aviv University